CLINICAL TRIAL: NCT06246227
Title: The Value of Circulating Tumour DNA in Early Detection of Recurrence of Melanoma
Brief Title: ctDNA for Early Detection of Recurrence in Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Danish Cancer Society (Other); Danish Cancer Research Foundation (Other); DCCC ctDNA Research Center (Unknown); CAG in Cancer immunotherapy (Unknown)
Responsible Party: Principal Investigator, Magnus Petur Bjarnason Obinah, Resident Medical Doctor, PhD Student, Herlev and Gentofte Hospital
Other Study IDs: H-18008586
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Melanoma
Keywords: ctDNA; Melanoma; Recurrence; Detection; ddPCR; NGS
MeSH Terms: conditions — Melanoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples will be analyzed for mutations using NGS Plasma harvested from collected blood samples, for later ddPCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Risk Melanoma Patients: Patients followed-up for Melanoma, Clinical Stages IIB - III and Resected Stage IV

SUMMARY:
This study examines circulating tumor DNA (ctDNA) as a biomarker for early detection of recurrence in high-risk patients, following treatment of primary melanoma. The hypothesis is that ctDNA can provide accurate detection of recurrence or metastasis, at the time of or earlier than current methods, leading to improved management and hopefully prognosis, based on earlier detection.

DETAILED DESCRIPTION:
This prospective, single-institution study will recruit patients attending follow-up for primary melanoma with high risk of recurrence, at the department of Plastic and Reconstructive Surgery, Herlev and Gentofte University Hospital, Copenhagen University.

Enrolled patients will undergo regular blood sampling. Samples will be centrifuged and plasma will be harvested and stored. In cases of metastasis or recurrence, tumor tissue samples will be analyzed using NGS to determine their mutational profile. Plasma samples will be analyzed for ctDNA corresponding to identified mutations. If ctDNA is detected, previous samples will be analyzed in reverse sequential order, until no ctDNA is detected.

Follow-up time after inclusion is five years or end of clinical-follow up, with an interim sample and data analysis scheduled for 2024 and final analysis scheduled for 2027-2028.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up for Primary Melanoma, Stages IIB to III and Resected Stage IV

Exclusion Criteria:

* Pregnancy
* Previous history of melanoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients followed for high-risk of recurrence, at the department of Plastic and Reconstructive Surgery, Herlev and Gentofte University Hospital, in the inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ctDNA for detection of metastatic disease | From enrollment to end of 5-year follow-up
  By analyzing blood samples of patients diagnosed with recurrence, we will establish the ability of ctDNA to detect known recurrence, and therefore be able to establish the sensitivity of the method.
Specificity of ctDNA for detection of metastatic disease | From enrollment to end of 5-year follow-up
  By assuming no ctDNA in healthy individuals and analyzing WBC from buffy-coat to correct for wild-type mutated DNA due to CHIP, we will be able to establish the specificity of the method.

SECONDARY OUTCOMES:
Time from detectable ctDNA to clinical og radiological suspicion of recurrence | From enrollment to end of 5-year follow-up
  We will start by analyzing the closest sample to the original suspicion of recurrence. In the event of ctDNA detection, previous samples will be analyzed in reverse sequential order, until no ctDNA is detected. This will allow us to establish a temporal relationship between the ability of ctDNA to detect recurrence and current surveillance methods.
Associations between ctDNA detection and quantification, and other biomarkers, including LDH, WBC differential, and HS-CRP | From enrollment to end of 5-year follow-up
  By measuring LDH, WBC Diff. and HS-CRP at every sampling, we will be able to establish the correlation between these currently accepted biomarkers for melanoma-specific survival and ctDNA measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet R Hölmich, MD, DMSc, Clinical Professor, Study Director — Dept. of Plastic and Reconstructive Surgery, Herlev and Gentofte University Hospital
Locations (1):
- Detp. of Pastic and Reconstructive Surgery, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No